CLINICAL TRIAL: NCT04389619
Title: Effect of Fractional Microneedling Radiofrequency Versus Intralesional Steroid Injection With and Without Microneedling on Tissue Levels of PDGF & CTGF in Hypertrophic Scars: a Randomized Comparative Clinical Trial.
Brief Title: Fractional Microneedling RF vs Intralesional Steroid With & Without Microneedling in Hypertrophic Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dermatology 13
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Hypertrophic Scars
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional Microneedling Radiofrequency (Experimental): In every patient, each one of the two scars, or each side of a large scar will be assigned to fractional microneedling radiofrequency parameters; Power: 6 v, Exposure time: 800 ms. Depth: 2.5 mm (using non-insulated micro-needles), Frequency: 2 Hz for 5 treatment sessions 4 weeks apart.
  Interventions: Device: Fractional Microneedling Radiofrequency
- Intralesional Steroid Injection with and without Microneedling (Active Comparator): In every patient, each one of the two scars, or the other side of a large scar will be assigned to intralesional steroids injection, Triamcinolone acetonide will be injected in concentration 1:2 (20 mg/dl) using insulin syringe. Microneedling will be done using the same tip of the fractional microneedling radiofrequency at same depth. Patients will receive 5 treatment sessions 4 weeks apart.
  Interventions: Procedure: Intralesional Steroid Injection with and without Microneedling

INTERVENTIONS:
Device: Fractional Microneedling Radiofrequency — In every patient, each one of the two scars, or each side of a large scar will be assigned to fractional microneedling radiofrequency. Fractional microneedling radiofrequency parameters; Power: 6 v, Exposure time: 800 ms. Depth: 2.5 mm (using non-insulated micro-needles), Frequency: 2 Hz for 5 treatment sessions 4 weeks apart.
  Arms: Fractional Microneedling Radiofrequency
Procedure: Intralesional Steroid Injection with and without Microneedling — In every patient, each one of the two scars, or the other side of a large scar will be assigned to intralesional steroids injection, Triamcinolone acetonide will be injected in concentration 1:2 (20 mg/dl) using insulin syringe. o Scars treated with intralesional steroids will be subgrouped into two groups, one group treated with only intralesional steroids and the other group treated with intralesional steroids and followed by microneedling. Microneedling will be done using the same tip of the fractional microneedling radiofrequency at same depth. Patients will receive 5 treatment sessions 4 weeks apart.
  Arms: Intralesional Steroid Injection with and without Microneedling

SUMMARY:
Comparing between the effect of Fractional Microneedling Radiofrequency Versus Intralesional Steroid Injection with and without Microneedling on Tissue levels of PDGF & CTGF in Hypertrophic Scars

DETAILED DESCRIPTION:
In each patient, each one of the two scars, or each side of a large scar will be assigned to one of the following treatment methods: 1-Fractional microneedling radiofrequency 2-Intralesional steroids injection. Scars treated with intralesional steroids will be subgrouped into two groups, one group treated with only intralesional steroids and the other group treated with intralesional steroids and followed by microneedling. Fractional microneedling radiofrequency parameters; Power: 6 v, Exposure time: 800 ms. Depth: 2.5 mm (using non-insulated micro-needles), Frequency: 2 Hz. For intralesional steroids injection, Triamcinolone acetonide will be injected in concentration 1:2 (20 mg/dl) using insulin syringe. Microneedling will be done using the same tip of the fractional microneedling radiofrequency at same depth. All patients will receive 5 treatment sessions 4 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mature hypertrophic scars.
* Patients with age above 18 years.
* Both males and females.
* Patients with two separate lesions, each 3 cm length at least OR a large sized lesion 10 cm length at least.

Exclusion Criteria:

* Patients with unrealistic expectations.
* Patients with active skin infections or autoimmune diseases.
* Non-compliant patients.
* Patients who had received any form of treatment for scars during the last six months.
* Recent use of isotretinoin within six months prior to the procedures.
* Patient with known allergy to lidocaine.
* Pregnancy & Lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Calculation of patient and observer scar assessment scale (POSAS) to assess change of hyertrophic scars | 6 months
  Calculation of patient and observer scar assessment scale (POSAS) before every session and one month after the last session to clinically assess change of hyertrophic scars
Photographic documentation will be performed to assess change of hypertrophic scar(s) | 6 months
  Photographic documentation will be performed by obtaining digital photographs for hypertrophic scar(s) before every session and one month after the last session.
Measurement of tissue levels of both platelet derived growth factor (PDGF) & connective tissue growth factor (CTGF) to assess change of hypertrophic scars | 6 months
  Measurement of tissue levels of both PDGF & CTGF to assess change of hypertrophic scars. Tissue levels of both PDGF & CTGF will be measured by PCR in biopsies obtained from the scar areas before the treatment sessions and one month after the last session

CONTACTS AND LOCATIONS:
Locations (1):
- Maha Fathy Elmasry, Cairo, Egypt